CLINICAL TRIAL: NCT05624294
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single Ascending Does/ Mulelple Ascending Does Study of CS0159 to Evaluate the Safety, Tolerability, Pharmacokynetics, and Food Effect in Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of CS0159 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0159-001A
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2mg CS0159 (Experimental): One tablet daily for seven days.
  Interventions: Drug: CS0159; Drug: Placebo
- 4mg CS0159 (Experimental): Two tablet daily for seven days.
  Interventions: Drug: CS0159; Drug: Placebo
- 6mg CS0159 (Experimental): Three tablet daily for seven days.
  Interventions: Drug: CS0159; Drug: Placebo

INTERVENTIONS:
Drug: CS0159 — Tablets administered orally
Drug: Placebo — Tablets administered orally

SUMMARY:
This is a phase I clinical bridging trial, randomized, double-blind, placebo-controlled, single ascending does/ mulelple ascending does study of CS0159 to evaluate the safety, tolerability, pharmacokynetics, pharmacodynamices, and food effect in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects of 18 years to 55 years.
2. Weight: Male≥50kg, female≥45kg BMI: 18~32kg/m².
3. In good health, determined by having no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluation.
4. Subject signs IFC and dates and subject must understand and follow test procedures and restrictions.

Exclusion Criteria:

1. Subjects with special dietary requirements and cannot follow a uniform diet.
2. Pregnant or nursing females or females who have pregnancy plans during the trial or within 3 months after the trial.
3. Any subject with SARS-CoV-2 infection, based on a positive polymerase chain reaction for SARS-CoV-2.
4. History or evidence of clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluations, procedures, or completion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events [Safety and Tolerability] | Upto day 15
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE) resulting in treatment discontinuation, and AE of special interest, from baseline up to 15 days.
Dose PK Parameter(C-max) | day 1, day 7
  Evaluate the Peak Plasma Concentration.
Dose PK Parameter(AUC) | day 1, day 7
  Evaluate the Area under the plasma concentration versus time curve.

SECONDARY OUTCOMES:
Food effect PK Parameter(C-max) | day 10
  Evaluate the Peak Plasma Concentration.
Food effect PK Parameter(AUC) | day 10
  Evaluate the Area under the plasma concentration versus time curve.
QTc analysis | day 1, day 7
  analysize the plasma Concentration relevance to QTcF

CONTACTS AND LOCATIONS:
Overall Officials: Yun Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No